CLINICAL TRIAL: NCT06964555
Title: Effect of Intravenous Low-Dose Ketamine Infusion With Intravenous Lignocaine Infusion on Post-Operative Pain in Patients Undergoing Laparoscopic Choleysystectomy Under General Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fazaia Ruth Pfau Medical College (Other)
Responsible Party: Principal Investigator, Syeda Hajrah Rehman, Principal Investigator, Fazaia Ruth Pfau Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FRPMC-IRB-2024-41
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Cholelithiases
Keywords: Cholelithiases; Cholecystectomy; Laparoscopy
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group L (Active Comparator): Just before the skin incision intravenous lignocaine was given.
  Interventions: Drug: Intravenous lignocaine
- Group K (Experimental): Just before the skin incision, intravenous ketamine was given
  Interventions: Drug: Intravenous Ketamine Infusions

INTERVENTIONS:
Drug: Intravenous Ketamine Infusions — Ketamine group received ketamine at 0.2mg/kg bolus intravenously followed by ketamine infusion at rate of 0.2mg/kg/hr throughout the surgery.
  Arms: Group K
Drug: Intravenous lignocaine — IV Lignocaine was given at the rate of 1 mg/kg/hr.
  Arms: Group L

SUMMARY:
Objective: To determine the effect of low-dose ketamine versus lignocaine on post-operative pain in patients undergoing LC under general anesthesia in a tertiary care hospital.

Sample Selection: Patients of both the gender of age at least 18 years, planned for elective LC with ASA grade I-II were included. Patients with obesity, history of alcohol consumptions, drug abusers, uncontrolled hypertension and diabetics, with chronic pain, allergic to study drugs, having neurological disorders, unable to understand pain scoring system and converted to open LC were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both the gender of age at least 18 years
* Patients planned for elective LC
* Patients with ASA grade I-II were included.

Exclusion Criteria:

* Patients with obesity,
* Patients with history of alcohol consumptions, uncontrolled hypertension and diabetics,
* Drug abusers
* Patients with chronic pain
* Patients allergic to study drugs
* Patients having neurological disorders or unable to understand pain scoring system
* Patients converted to open LC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Post operative Pain | 24 hours
  Pain was assessed using Numeric Rating Scale which is a ten point scoring scale ranging from 0-10 for ranking pain where 0 means no and 10 means worst pain.

SECONDARY OUTCOMES:
Time to rescue analgesia | 24 hours
  Time to rescue analgesia was defined as time point at which patient will be given first rescue analgesia for pain of score more 5 or above.
Wound Closure | End of Surgery
  The time between the incision and the wound's closure was used to define the length of the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Fazaia Ruth Pfau Medical College, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No